CLINICAL TRIAL: NCT06981039
Title: The WASP Trial (Wiring Versus Anterior Star Plate): Comparison of Patella Plating Versus Tension Band Wiring for the Treatment of Unstable Patellar Fractures: A Randomized Controlled Trial
Brief Title: Comparison of Patella Plating Versus Tension Band Wiring for the Treatment of Unstable Patellar Fractures
Acronym: WASP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Christian Xinshuo Fang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 24-025
Record Dates: First submitted 2025-05-02; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Patella Fracture
Keywords: trauma; knee injury; Tension Band Wiring; Patella fracture; Anatomical locking plate fixation
MeSH Terms: conditions — Patella Fracture; Wounds and Injuries; Knee Injuries

STUDY DESIGN:
Intervention Model Description: Pragmatic, double-blind randomized controlled trial with 60 patients in two interventional arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomly assigned to either one of the interventional arms and will not be informed of the randomization result.
  A blinded reviewer will assess the radiographs, surgical quality, and clinical outcomes postoperatively and during study follow-ups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patella Anatomical Locking Plate Group (Anterior Star Plate) (Experimental): Fracture repair surgery using the patella anatomical locking plate
  Interventions: Device: Patella Anatomical Locking Plate
- Tension Band Wiring Group (Wiring) (Active Comparator): Fracture repair surgery with a tension band wire construct
  Interventions: Device: Tension Band Wiring

INTERVENTIONS:
Device: Patella Anatomical Locking Plate — Patients in the patella anatomical locking plate group will undergo internal fixation with an anterior locking plate and screw construct using the 2.7mm variable angle (VA) locking patella plating system (DePuy Synthes, Zuchwil, Switzerland)
  Arms: Patella Anatomical Locking Plate Group (Anterior Star Plate)
Device: Tension Band Wiring — Patients in the tension band wiring group will undergo open anatomical reduction and internal fixation with a tension band wire construct.
  Arms: Tension Band Wiring Group (Wiring)

SUMMARY:
This study aims to compare the efficacy and safety of patella anatomical locking plate fixation versus tension band wiring in the treatment of patellar fractures.

DETAILED DESCRIPTION:
Patellar fractures are a common injury that can cause significant pain and disability. Conventional treatment options frequently include tension band wiring (TBW) with or without axial K-Wires or through cannulated screws. However, tension band wiring does have its issues, including implant prominence and frequent reoperation rates, especially for comminuted patella fractures.

More recently, plate fixation has become increasingly more prevalent in the past decade. Initially, this began with small fragment or mini-fragment plates; which progressed to mesh locking plates and now, anatomical locking patella plates. Biomechanical studies have shown greater loads to failure, less fracture gapping or fracture displacement with locking plate fixation compared to TBW. Its low profile construct and round edges may be more tolerable to patients and less prominent than TBW. Furthermore, another possible advantage of plate fixation is the avoidance of quadricep and patellar tendon insertion scarring, as they do not need to be dissected or passed through for fixation as in TBW. This is the first randomized controlled trial comparing anatomical locking plate fixation and conventional tension band wiring for patella fractures to be performed. This study aims to compare the efficacy and safety of these two methods in the treatment of patellar fractures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Diagnosed with an isolated closed injury, displaced, unstable fracture with displacement >2mm (AO/OTA Classification 34-B and C with surgical indication)
* Able to give consent

Exclusion Criteria:

* History of previous knee surgery
* Poly trauma,
* Ongoing malignancy
* Pre-existing severe knee osteoarthritis (>KL stage 4)
* Stroke
* Other neurological conditions/injuries to the lower limb
* Unfit for surgical anaesthesia
* Non-ambulatory
* Unable to consent or follow commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Region specific patient reported functional outcome scores - Knee Injury and Osteoarthritis Outcome Score (KOOS) | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used, and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems), and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Tegner Lysholm Knee Score | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  The Lysholm Knee Score calculates and grades an overall score from 0 to 100 based on 8 domains: squatting, locking, pain, stair climbing, support, instability, and edema. Scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.
Tegner Activity Scale | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  The Tegner Activity Scale is a one-item questionnaire that is scored on an 11-item scale (0 to 10) based on the patient's reported level of activity/work. A level of 0 represents maximum disability while a level of 10 represents elite sports athletes. Patients are asked to choose the highest level of activity they partake in at that moment.

SECONDARY OUTCOMES:
Radiographic outcomes | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Subjects' X-rays will be assessed for fracture healing progress.
Incidence of Complications | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Complications such as fracture site infection, implant failure, and re-operation will be assessed and recorded
Subjective Implant Impingement Questionnaire | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  The questionnaire consists of 11 questions assessing the level of implant impingement reported by the patient, with a final score ranging from 0 (no impingement) to 20 (consistent impingement).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fang, Principal Investigator — Dept of Orthopaedics and Traumatology, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset to be included as supplementary data in final publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of study completion
Access Criteria: Additional information available upon reasonable request of principal investigator